CLINICAL TRIAL: NCT03807089
Title: Adenoma Detection Rate With a New Pediatric Colonoscope With a Short Turn Radius (Pentax Retroview) Compared With a Standard Pentax Pediatric Colonoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pentax Medical (Industry)
Responsible Party: Principal Investigator, Norman Nishioka, MD, Director of Endoscopy, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014P000677
Record Dates: First submitted 2019-01-11; First posted 2019-01-16 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; colon cancer screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Short-Turn Radius Colonoscope (Experimental): Colonoscopy performed with Short-Turn Radius Colonoscope. The colonoscope will provide a forward-facing view of the colon during advancement to the cecum (standard of care). The scope will then be withdrawn all the way to the rectum and the colon will be inspected using the forward-facing view (standard of care). The colonoscope will then be re-advanced to the cecum and be withdrawn using the retrograde view.
  Interventions: Device: Short-Turn Radius Colonoscope
- Conventional Pediatric Colonoscope (Active Comparator): Colonoscopy will be performed with a conventional pediatric colonoscope. During withdrawal, the colon will be inspected using the forward-facing view (standard of care). The colonoscope will then be re-advanced to the cecum and again withdrawn using the forward-facing view.
  Interventions: Device: Conventional Pediatric Colonoscope

INTERVENTIONS:
Device: Conventional Pediatric Colonoscope
  Other Names: Pentax Model EG-2490K
  Arms: Conventional Pediatric Colonoscope
Device: Short-Turn Radius Colonoscope
  Other Names: Pentax Model EC-3490TLi
  Arms: Short-Turn Radius Colonoscope

SUMMARY:
The purpose of this study is to determine whether the new colonoscope that provides both a traditional and a retrograde view (bending 180 degrees to look behind itself) of the colon can detect more polyps than a standard colonoscope that only provides a forward-facing view. The investigators wish to effectively demonstrate the utility of the new colonoscope (Pentax Retroview Colonoscope) as the objective of this study is to determine polyp and adenoma detection rates in human subjects undergoing colonoscopy for polyp surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide Informed Consent
* Age > 40
* Surveillance Colonoscopy (History of Adenomas)

Exclusion Criteria:

* Poor or Fair Bowel Prep
* Difficult First Insertion
* Familial Polyposis
* Inflammatory Bowel Disease
* Pregnancy
* Active GI Bleeding
* Prior colonic or rectal resection
* Conserved Sattus
* Colonoscopy less than 3 years ago
* Screening Colonoscopy
* Colonoscopy done to evaluate systems like abdominal pain, diarrhea, constipation, change in bowel habits

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman S Nishioka, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Cutler CS, Lemmel GT, Rahmani EY, Clark DW, Helper DJ, Lehman GA, Mark DG. Colonoscopic miss rates of adenomas determined by back-to-back colonoscopies. Gastroenterology. 1997 Jan;112(1):24-8. doi: 10.1016/s0016-5085(97)70214-2. PMID 8978338
- [Background] Rex DK, Rahmani EY, Haseman JH, Lemmel GT, Kaster S, Buckley JS. Relative sensitivity of colonoscopy and barium enema for detection of colorectal cancer in clinical practice. Gastroenterology. 1997 Jan;112(1):17-23. doi: 10.1016/s0016-5085(97)70213-0. PMID 8978337
- [Background] Baxter NN, Goldwasser MA, Paszat LF, Saskin R, Urbach DR, Rabeneck L. Association of colonoscopy and death from colorectal cancer. Ann Intern Med. 2009 Jan 6;150(1):1-8. doi: 10.7326/0003-4819-150-1-200901060-00306. Epub 2008 Dec 15. PMID 19075198
- [Background] DeMarco DC, Odstrcil E, Lara LF, Bass D, Herdman C, Kinney T, Gupta K, Wolf L, Dewar T, Deas TM, Mehta MK, Anwer MB, Pellish R, Hamilton JK, Polter D, Reddy KG, Hanan I. Impact of experience with a retrograde-viewing device on adenoma detection rates and withdrawal times during colonoscopy: the Third Eye Retroscope study group. Gastrointest Endosc. 2010 Mar;71(3):542-50. doi: 10.1016/j.gie.2009.12.021. PMID 20189513
- [Background] Kessler WR, Rex DK. Impact of bending section length on insertion and retroflexion properties of pediatric and adult colonoscopes. Am J Gastroenterol. 2005 Jun;100(6):1290-5. doi: 10.1111/j.1572-0241.2005.41454.x. PMID 15929759
- [Background] Waye JD, Heigh RI, Fleischer DE, Leighton JA, Gurudu S, Aldrich LB, Li J, Ramrakhiani S, Edmundowicz SA, Early DS, Jonnalagadda S, Bresalier RS, Kessler WR, Rex DK. A retrograde-viewing device improves detection of adenomas in the colon: a prospective efficacy evaluation (with videos). Gastrointest Endosc. 2010 Mar;71(3):551-6. doi: 10.1016/j.gie.2009.09.043. Epub 2009 Dec 16. PMID 20018280

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 89 subjects were excluded (poor bowel preparation [n = 45], prior colonic resection [n = 3], difficult first insertion [n=45], not over 40 [n = 1], no history of adenomatous colorectal polyps [n = 1], device related reasons [n = 1])
Groups:
- Short-Turn Radius Colonoscope: Colonoscopy performed with Short-Turn Radius Colonoscope. The colonoscope will provide a forward-facing view of the colon during advancement to the cecum (standard of care). The scope will then be withdrawn all the way to the rectum and the colon will be inspected using the forward-facing view (standard of care). The colonoscope will then be re-advanced to the cecum and be withdrawn using the retrograde view.
  Short-Turn Radius Colonoscope
- Conventional Pediatric Colonoscope: Colonoscopy will be performed with a conventional pediatric colonoscope. During withdrawal, the colon will be inspected using the forward-facing view (standard of care). The colonoscope will then be re-advanced to the cecum and again withdrawn using the forward-facing view.
  Conventional Pediatric Colonoscope
Period: Overall Study
Arm/Group | Short-Turn Radius Colonoscope | Conventional Pediatric Colonoscope
Started | 101 | 93
Completed | 101 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short-Turn Radius Colonoscope | Conventional Pediatric Colonoscope | Total
Number analyzed (Participants) | 101 | 93 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.13) | 65.8 (8.38) | 65.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 59 | 118
  Male | 42 | 34 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 101 | 93 | 194

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With At Least One Adenoma
Description: Compare adenoma detection rate between patients undergoing a colonoscopy with Pentax Retroview colonoscope and pediatric colonoscope.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Short-Turn Radius Colonoscope | Conventional Pediatric Colonoscope
Number analyzed (Participants) | 101 | 93
Participants | 63 | 68

2. Secondary Outcome: Overall Polyp Detection Rate
Description: Compare polyp detection rate (percent of patients with at least one polyp detected) between patients undergoing a colonoscopy with Pentax Retroview colonoscope and pediatric colonoscope.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Short-Turn Radius Colonoscope | Conventional Pediatric Colonoscope
Number analyzed (Participants) | 101 | 93
Participants | 72 | 78

3. Secondary Outcome: Mean Number of Adenomas Identified Per Patient With Polyps
Description: Compare average number of adenomas found per patient with polyps between patients undergoing a colonoscopy with Pentax Retroview colonoscope and pediatric colonoscope.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: Number of Adenomas Per Patient
Arm/Group | Short-Turn Radius Colonoscope | Conventional Pediatric Colonoscope
Number analyzed (Participants) | 101 | 93
Number of Adenomas Per Patient | 2.48 (2.05) | 2.50 (1.56)

4. Other Pre Specified Outcome: Size of Polyps Detected
Description: Polyp size was estimated prior to polypectomy by comparing the polyp with objects of known dimension (biopsy forceps, polypectomy snares).
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Short-Turn Radius Colonoscope | Conventional Pediatric Colonoscope
Number analyzed (Participants) | 101 | 93
mm | 4.89 (2.92) | 4.50 (2.30)

5. Other Pre Specified Outcome: Size of Adenomas Detected
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Short-Turn Radius Colonoscope | Conventional Pediatric Colonoscope
Number analyzed (Participants) | 101 | 93
mm | 5.15 (3.04) | 4.69 (2.40)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected during the procedure, an average of 1 hour.
Arm/Group | Short-Turn Radius Colonoscope | Conventional Pediatric Colonoscope
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/93
Other Adverse Events (participants affected / at risk) | 0/101 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT03807089/Prot_SAP_001.pdf